CLINICAL TRIAL: NCT05081856
Title: The Effect of Modular Carrying System on Patient Outcomes in the Mobilization of Patients With a Chest Tube
Brief Title: Use Modular Medical Equipment Vehicle in Mobilization of Patient With Chest Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, pınar dogan, Asst.Prof., Istanbul Medipol University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 12093487
Record Dates: First submitted 2021-08-16; First posted 2021-10-18 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Mobility Limitation; Sleep Quality; Pain; Comfort; Time of the Removal Chest Tube
Keywords: care outcomes; mobilization; chest tube
MeSH Terms: conditions — Mobility Limitation; Sleep Initiation and Maintenance Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Interventional study with posttest control group
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The group mobilized for at least 20 minutes 6 times a day with a modular medical equipment carrying vehicle
  Interventions: Other: mobilization with moduler medical equipment carring vehicle
- control group (No Intervention): The group mobilized for at least 20 minutes 6 times a day with a routin practice

INTERVENTIONS:
Other: mobilization with moduler medical equipment carring vehicle — Mobilization of the patients was carried out with the vehicle in their modular vehicle.
  Arms: intervention group

SUMMARY:
in this study, it was aimed to examine the effect of the modular carrying system on the outcomes of care in the mobilization of patients with a chest tube. The population of the study consisted of patients followed in Yedikule Chest Diseases, and Thoracic Surgery Training and Research Hospital between October 2019 and January 2021, and the sample consisted of 83 patients who met the inclusion criteria. The study was performed with the intervention group (n=37) mobilized with the Modular medical equipment carrying vehicle and the control group (n=46) mobilized with the routine application.

DETAILED DESCRIPTION:
Within the scope of the study, a Modular medical equipment carrying vehicle was developed by the researchers to ensure the safe and comfortable mobilization of patients with chest tube and additional medical equipment. This vehicle has been designed to maintain the level of the chest tube during mobilization and to prevent it from tipping over.Patients in the intervention group were mobilized with the help of this Modular medical equipment carrying vehicle for 20 minutes at least 6 times a day. Patients in the control group were mobilized at least 6 times a day for 20 minutes with clinical routine practice.

ELIGIBILITY:
Inclusion Criteria:

* chest tube inserted due to open surgery, hemodynamically stable, followed up in the clinic for at least 5 days, first mobilized after chest tube inserted

Exclusion Criteria:

* have a mental or psychological illness, hemodynamically unstable

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
general comfort scale score | first day and fifth day
  monitoring of changes in the general comfort levels of the patients during the intervention
Richard Campell sleep quality scale score | every day for five days
  monitoring of changes in the sleep quality of the patients during the intervention
pain scale score | every day for five days
  monitoring of changes in the pain levels of the patients during the intervention
patient mobility scale score | every day for five days
  monitoring of changes in the mobility of the patients during the intervention
drain removal time (day (median)) | the day the drain was removed
  monitoring of changes in the drain removal time of the patients during the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Dogan, Asst.Prof., Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data from the study will be reported over the levels of change in maintenance results. The study report is aimed to be published as a clinical research report.
Supporting Information: CSR
Time Frame: Data will be used for 2 years
Access Criteria: increase in sleep, comfort and mobility level of patients mobilized with this tool, decrease in pain and drain removal time